CLINICAL TRIAL: NCT02500537
Title: A Post-market Study of the Endo GIA™ Reinforced Reload With Tri-Staple™ Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVRRBT0451
Record Dates: First submitted 2015-06-01; First posted 2015-07-16 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Non-emergent, Abdominal or Thoracic Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abdominal Procedures (Experimental): Abdominal procedures may include, but are not limited to, laparoscopic sleeve gastrectomy (LSG), laparoscopic Roux-en-Y gastric bypass (LRYGB), and biliopancreatic diversion, as well as hepatic and pancreatic resection.
  Device: Endo GIA™ Reinforced Reload with Tri-Staple™ Technology
  Interventions: Device: Endo GIA™ Reinforced Reload with Tri-Staple™ Technology
- Thoracic Procedures (Experimental): Thoracic procedures may include, but are not limited to wedge resection and lobectomy, and may include video assisted thoracic surgery (VATS) or open procedures.
  Device: Endo GIA™ Reinforced Reload with Tri-Staple™ Technology
  Interventions: Device: Endo GIA™ Reinforced Reload with Tri-Staple™ Technology

INTERVENTIONS:
Device: Endo GIA™ Reinforced Reload with Tri-Staple™ Technology — Endo GIA™ Reinforced Reload with Tri-Staple™ Technology (Universal Handle)

SUMMARY:
A post-market study of the Endo GIA™ Reinforced Reload with Tri-Staple™ Technology.

DETAILED DESCRIPTION:
The objective of this prospective, two-arm, multicenter, post-market study is to evaluate safety through the incidence of reported device-related adverse events (AEs) through 30 days following use of the Endo GIA™ Reinforced Reload with Tri-Staple™ Technology in subjects undergoing indicated abdominal or thoracic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be 18-80 years of age
2. The subject must be willing and able to participate in the study procedures and to understand and sign the informed consent
3. The subject is undergoing an indicated primary abdominal or thoracic procedure where the Endo GIA™ Reinforced Reload with Tri-Staple™ Technology (Universal Handle) will be used per its Instructions For Use (IFU)

   * Thoracic procedures may include, but are not limited to, wedge resection and lobectomy, and may include video assisted thoracic surgery (VATS) or open procedures.
   * Abdominal procedures may include, but are not limited to, laparoscopic sleeve gastrectomy (LSG), laparoscopic Roux-en-Y gastric bypass (LRYGB), and biliopancreatic diversion, as well as hepatic and pancreatic resection.
4. For thoracic subjects: the subject has a FEV1 ≥40%

Exclusion Criteria:

1. Subjects undergoing cardiac and vascular procedures
2. The procedure is an emergency procedure
3. The procedure is a revision/reoperation for the same indication
4. Any female subject who is pregnant

   a. Females of child-bearing potential will be required to provide either a urine pregnancy test or serum pregnancy test (except for subjects who are surgically sterile or are post-menopausal for at least two years)
5. Any subject who is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity)
6. The subject is unable or unwilling to comply with the study requirements or follow-up schedule
7. The subject has comorbidities which, in the opinion of the Investigator, will not be appropriate for the study or the subject has an estimated life expectancy of less than 6 months
8. The subject has been diagnosed with a bleeding disorder and/or is undergoing active and not reversed anticoagulant treatment
9. The subject is concurrently enrolled in an investigational drug or device research study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ahmed, PhD, FRCS, Principal Investigator — St Mary's Hospital, London
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Abdominal Procedures: Abdominal procedures may include, but are not limited to, laparoscopic sleeve gastrectomy (LSG), laparoscopic Roux-en-Y gastric bypass (LRYGB), and biliopancreatic diversion, as well as hepatic and pancreatic resection
  Endo GIA™ Reinforced Reload with Tri-Staple™ Technology: Endo GIA™ Reinforced Reload with Tri-Staple™ Technology (Universal Handle)
- Thoracic Procedures: Thoracic procedures may include, but are not limited to wedge resection and lobectomy, and may include video assisted thoracic surgery (VATS) or open procedures
  Endo GIA™ Reinforced Reload with Tri-Staple™ Technology: Endo GIA™ Reinforced Reload with Tri-Staple™ Technology (Universal Handle)
Period: Overall Study
Arm/Group | Abdominal Procedures | Thoracic Procedures
Started | 60 | 40
Completed | 57 | 39
Not Completed | 3 | 1
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdominal Procedures | Thoracic Procedures | Total
Number analyzed (Participants) | 60 | 40 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (13.56) | 64.6 (9.7) | 52.7 (15.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 20 | 61
  Male | 19 | 20 | 39
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 44.3 (7.06) | 27.9 (5.87) | 36.4 (10.73)
FEV1 Score (thoracic) [Mean (Standard Deviation); unit: percent] — Population: FEV1 Score is captured for the thoracic population
  percent
    number analyzed (Participants) | 0 | 40 | 40
    (all) |  | 82.2 (20.41) | 82.2 (20.41)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Incidence of Reported Device-related Adverse Events (AEs) Through 30 Days Following Indicated Abdominal or Thoracic Procedures.
Time Frame: Through 30 Days
Measure: Number; unit: Device related adverse events
Arm/Group | Abdominal Procedures | Thoracic Procedures
Number analyzed (Participants) | 60 | 40
Device related adverse events | 2 | 1

2. Secondary Outcome: Staple Line Assessment: Incidence of Staple Line Bleeding
Description: The incidence of staple line bleeding will be measured as ≥ 50 cc
Time Frame: Day 0
Measure: Number; unit: incidences of staple line bleeding
Arm/Group | Abdominal Procedures | Thoracic Procedures
Number analyzed (Participants) | 60 | 40
incidences of staple line bleeding | 0 | 0

3. Secondary Outcome: Staple Line Assessment: Incidence of Leakage
Description: As measured by air leak test, or standard of care, as applicable
Time Frame: Day 0
Measure: Number; unit: incidences of leakage
Arm/Group | Abdominal Procedures | Thoracic Procedures
Number analyzed (Participants) | 60 | 40
incidences of leakage | 0 | 3

4. Secondary Outcome: Staple Line Assessment: Duration of Leakage, Post-Op
Description: Duration of leakage based on chest tube drainage in days
Time Frame: Participants will be followed for the duration of hospital stay, on average up to 5 days
Population: Thoracic patients only
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Thoracic Procedures
Number analyzed (Participants) | 40
days | 7.7 (5.51)

5. Secondary Outcome: Staple Line Assessment: Incidence of Leakage; Post-Op
Description: The incidence of leakage for abdominal procedures; Post-up
Time Frame: Participants will be followed for the duration of hospital stay, on average up to 5 days
Population: Abdominal patients only
Measure: Number; unit: participants
Arm/Group | Abdominal Procedures
Number analyzed (Participants) | 60
participants | 1

6. Secondary Outcome: Staple Line Assessment: Incidence of Post-operative Infection
Description: Incidence of post-operative infection at the staple line in abdominal patients and thoracic patients
Time Frame: Participants will be followed for the duration of hospital stay, on average up to 5 days
Measure: Number; unit: participants
Arm/Group | Abdominal Procedures | Thoracic Procedures
Number analyzed (Participants) | 60 | 40
participants | 1 | 4

7. Secondary Outcome: Staple Line Assessment:
Description: Number of additional intervention(s) to treat staple-line failure
Time Frame: Participants will be followed for the duration of hospital stay, on average up to 5 days post-op
Measure: Number; unit: participants
Arm/Group | Abdominal Procedures | Thoracic Procedures
Number analyzed (Participants) | 60 | 40
participants | 2 | 0

8. Secondary Outcome: Incidence of Repeat Hospital Admissions for Procedural-related Complications
Description: Incidence of repeat hospital admissions for procedural-related complications for up to 30 days following procedure
Time Frame: 30 Days following procedure
Measure: Number; unit: participants
Arm/Group | Abdominal Procedures | Thoracic Procedures
Number analyzed (Participants) | 60 | 40
participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Abdominal Procedures | Thoracic Procedures
All-Cause Mortality (participants affected / at risk) | 2/60 | 0/40
Serious Adverse Events (participants affected / at risk) | 12/60 | 5/40
Other Adverse Events (participants affected / at risk) | 14/60 | 14/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abdominal Procedures (N=60) | Thoracic Procedures (N=40)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic rupture (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Complication of device removal (General disorders) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal Procedures (N=60) | Thoracic Procedures (N=40)
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 | 0
Confusion postoperative (Injury, poisoning and procedural complications) | 1 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 2
Incision site infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 2
Oxygen supplementation (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days